CLINICAL TRIAL: NCT03249610
Title: Worksite Intervention Trial With Multi-Component Lifestyle Intervention and Digital Health Platform for Reduction of Body Weight and Cardio-metabolic Risk Factors
Brief Title: Randomized Control Trial for Overweight Employees in Worksites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Sprim Advanced Life Sciences (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Dr Anoop Misra, Professor, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Worksite_2014
Record Dates: First submitted 2017-07-01; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome; Lifestyle Risk Reduction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Jindal Steel Pvt Ltd (Experimental): Lifestyle intervention given
  Interventions: Behavioral: Lifestyle intervention
- Maruti Udyog Ltd (Experimental): Lifestyle intervention given
  Interventions: Behavioral: Lifestyle intervention
- Tata Capital (No Intervention): Control arm so no intervention given
- Powergrid Corporation (No Intervention): Control arm so no intervention given

INTERVENTIONS:
Behavioral: Lifestyle intervention — Intervention Trial with Multi-Component Lifestyle Intervention for reduction of body weight and cardio-metabolic risk factors
  Arms: Jindal Steel Pvt Ltd; Maruti Udyog Ltd

SUMMARY:
Impact of lifestyle intervention in at-risk Asian Indians at worksite remains largely unexplored. The aim of this study was to assess impact of the multi-component interventions on body weight, body fat patterning and cardio-metabolic risk factors in overweight individuals working in corporate worksites in New Delhi, north India.

DETAILED DESCRIPTION:
A randomized open label clinical trial is planned in 4 worksites. The total study duration is 18 months. Four workplace sites will be divided into two active intervention and two control sites. Intensive awareness generation activities for overweight and obese employees and a general awareness health, nutrition and physical education programme for the rest of the employees. The study subjects will be part of awareness sessions which will be conducted in the 6 month intervention period. Besides group sessions individual diet charts will also be worked out by a trained nutritionist. Physical activity advice will be provided to them keeping their specific requirements in mind. Pedometers will be provided to them and they will be encouraged to walk for 15 minutes in pre-lunch period. Leg movements at the desk will also be encouraged.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (≥23kg/m 2 ) individuals in the age group 25-55 years
* Individuals who are willing to participate in the study

Exclusion Criteria:

* Previously diagnosed diabetics and patients with coronary artery disease.
* Have received any medication within last one month which could potentially influence insulin secretion, insulin sensitivity, (e.g. metformin, thiazolidinediones, steroids etc.) and on any medication that activate steroid and xenobiotic receptors
* Pregnant and lactating women
* Severe end organ damage or chronic diseases:renal/hepatic failure, any malignancy, major systemic illness etc.
* Known case of HIV infection
* Unwillingness to participate in the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2017-03-12 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects with reduced Body Mass Index | 6 months
  Body Mass Index measured in kg/m^2

SECONDARY OUTCOMES:
Number of subjects with reduced Fasting Blood Glucose | 6 months
  Fasting Blood Glucose measured in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anoop Misra, Principal Investigator — Diabetes Foundation, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shrivastava U, Fatma M, Mohan S, Singh P, Misra A. Randomized Control Trial for Reduction of Body Weight, Body Fat Patterning, and Cardiometabolic Risk Factors in Overweight Worksite Employees in Delhi, India. J Diabetes Res. 2017;2017:7254174. doi: 10.1155/2017/7254174. Epub 2017 Nov 29. PMID 29318159